CLINICAL TRIAL: NCT02458989
Title: A Randomized Controlled Trial Comparing The Cosmetic Outcome Of Electrocautery Versus Scalpel For Thyroidectomy Incisions
Brief Title: Thyroid Cosmesis Study at St. Paul's Hospital, Vancouver BC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Sam M. Wiseman (Other)
Responsible Party: Sponsor-Investigator, Dr. Sam M. Wiseman, Principal Investigator, St. Paul's Hospital, Canada
Organization: St. Paul's Hospital, Canada (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Thyroid Cosmesis H14-02408
Record Dates: First submitted 2015-03-19; First posted 2015-06-01 (Estimated); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Surgery
Keywords: Thyroidectomy; Thyroid surgery; Scalpel; Electrocautery
MeSH Terms: interventions — Laser Therapy; Electrocoagulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Scalpel (Active Comparator): Use of a scalpel as a first incision during thyroid operation.
  Interventions: Procedure: Scalpel
- Electrocautery (Experimental): Use of an electrocautery as a first incision during thyroid operation.
  Interventions: Procedure: Electrocautery

INTERVENTIONS:
Procedure: Scalpel — Use of a scalpel as a first incision during thyroid operation
  Arms: Scalpel
Procedure: Electrocautery — Use of an electrocautery as a first incision during thyroid operation
  Arms: Electrocautery

SUMMARY:
This study looks at the difference in surgical scar outcomes between two different surgical incision methods during thyroid surgery: scalpel vs electrocautery. Patients who are already scheduled for thyroid surgery with Dr. Sam Wiseman, Endocrine Surgeon at St. Paul's Hospital, and that meet the eligibility criteria for this study will be invited to participate. After signing the informed consent form, participants will be randomized into either one of the two incision methods, but will not know which one they receive. There will be two follow-up time points: one at 6 and another at 12 months post-operative. At these time points the research team will send a letter to the participant asking them to rate the appearance of their surgical scar. They will also be asked to take a picture of their scar and send it back to the research team, so that the research team can make an assessment of their surgical scar. The study concludes when the 12 month follow-up is complete.

DETAILED DESCRIPTION:
Purpose:

To evaluates the difference in thyroid cosmesis between two different surgical incision methods during thyroidectomy: scalpel vs electrocautery.

Hypotheses:

The investigators' hypotheses is that there is no difference in the cosmetic outcome of surgical incision during thyroidectomy by either a scalpel or electrocautery.

Justification:

Very few studies have addressed whether electrocautery produces a cosmetically inferior surgical scar in an objective manner. While some studies have commented briefly on the cosmesis of electrocautery scars, only one previous randomized clinical trials to date have evaluated the cosmesis of electrocautery and scalpel incisions using a validated scar assessment tool. In this study, Chau et al. found that after 6 months postoperatively there was no difference in objective cosmetic outcome or subjective patient satisfaction between the two techniques. This study was a relatively smaller trial, evaluating a total of 38 incisions, thus a larger scale study would be warranted.

A further advantage of electrocautery over scalpels is the decreased risk of surgical injuries. Approximately 17% of all surgical sharps injuries are due to scalpel blades, while only 2% were associated with electrocautery devices. As awareness and concern over blood born diseases increases, further efforts to reduce sharp injuries including replacing scalpels with electrocautery when possible should be investigated.

Objectives:

Aim 1: To compare the cosmetic outcome of surgical scars resulting from scalpel and electrocautery incisions.

Aim 2: To determine rates of wound infection associated with each technique.

Aim 3: To assess if electrocautery incisions are associated with a difference in postoperative pain compared to incisions made by a scalpel.

Research Method:

Patients who are already scheduled for thyroid surgery with Dr. Sam Wiseman at St. Paul's Hospital in Vancouver, BC, and that meet the eligibility criteria for this study will be invited to participate. After signing the informed consent form, participants will be randomized into either one of the two incision methods, but will be blinded as to which one they receive. There will be two follow-up time points: one at 6 months and another at 12 months postoperative. At these time points the research team will send a letter to the participant asking them to rate the appearance of their surgical scar, rate of their wound infection and the degree of their post operative pain using the Patient Observer Scar Assessment Scale (POSAS). They will also be asked to take a picture of their scar and send it back to the research team so the research team can make a similar assessment.

Statistical Analysis:

Once the research team receives the participant's questionnaire and photo, the images of their surgical scars will be evaluated by independent, trained, and blinded observers who will use the Patient Observer Scar Assessment Scale (POSAS) and the Vancouver Scar Scale (VSS) to evaluate the cosmesis of the surgical scar. The participants questionnaires will also be evaluated by the surgical team to assess Objective: Aim #3. The study concludes when the 12 month follow-up and these assessment by the research team is complete.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old who have consented to conventional thyroid surgery with Dr. Sam Wiseman at St Paul's Hospital (Vancouver, BC) will be asked to participate.

Exclusion Criteria:

* Patients will be excluded if they have had prior surgical incisions at the site of expected surgical incision, connective tissue disorders (e.g. Ehrlos Danlos syndrome), known keloid predilection, and lack of informed consent.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-03; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Appearance of surgical scar | 6 months post operative
Appearance of surgical scar | 12 months post operative

SECONDARY OUTCOMES:
Rate of wound infection | 6 months post operative
Rate of wound infection | 12 months post operative

OTHER OUTCOMES:
Scar pain score on the POSAS Patient Scale | 6 months post operative
Scar pain score on the POSAS Patient Scale | 12 months post operative

CONTACTS AND LOCATIONS:
Overall Officials: Sam M Wiseman, MD, Principal Investigator — University of British Columbia and St. Paul's Hospital
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Chau JK, Dzigielewski P, Mlynarek A, Cote DW, Allen H, Harris JR, Seikaly HR. Steel scalpel versus electrocautery blade: comparison of cosmetic and patient satisfaction outcomes of different incision methods. J Otolaryngol Head Neck Surg. 2009 Aug;38(4):427-33. PMID 19755082